CLINICAL TRIAL: NCT04194450
Title: The Effect of Acute Exogenous Oral Ketone Supplementation on Blood Glucose Levels in Type 2 Diabetes
Brief Title: Exogenous Ketones in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H19-02947
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Results first posted 2023-12-11 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Ketosis; Type 2 Diabetes
MeSH Terms: conditions — Ketosis; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Placebo masked with flavouring and participants consume in opaque containers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone monoester (Experimental): Acute dose of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate (0.3 g/kg body weight)
  Interventions: Dietary Supplement: Ketone monoester
- Placebo (Placebo Comparator): Acute dose of flavour-matched placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone monoester — Acute ingestion of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate prior to assessment of outcomes.
  Arms: Ketone monoester
Dietary Supplement: Placebo — Acute ingestion of taste-matched placebo prior to assessment of outcomes.
  Arms: Placebo

SUMMARY:
Exogenous ketone supplements are proposed to have glucose-lowering potential, provide an alternative fuel for the brain and to enhance cognitive function. No studies have tested whether exogenous ketones can lower blood glucose in people with type 2 diabetes. In addition, the impact of exogenous ketones on brain blood flow, cognitive function or brain-derived neurotrophic factor in humans is unknown. The purpose of this study is to determine if acutely ingesting exogenous ketones, in the form of a ketone monoester drink, can lower glucose and improve measures of brain/cognitive function in humans with type 2 diabetes. Participants will consume a ketone monoester drink or placebo with blood samples, brain blood flow, and cognitive function assessed over 180 minutes. The researchers will also test how the ketone monoester drink impacts appetite and measures of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* physician-diagnosed type 2 diabetes of ≥1 year
* current hemoglobin A1C (HbA1c) of 6.5-8.0%
* treatment with lifestyle or stable (≥3 months) oral glucose-lowering medications
* blood pressure of <160/99 mm Hg assessed according to guidelines
* non-smoking
* no prior history of cardiovascular disease or stroke
* not on hormone replacement therapy, corticosteroids, or anti-inflammatory medications
* 20-75 years old

Exclusion Criteria:

* being a competitive endurance athlete
* taking exogenous insulin or sodium glucose transporter 2 (SGLT2) inhibitors
* following a ketogenic diet, low-calorie diet, periodic fasting regimen, or consume ketogenic supplements
* being unable to travel to and from the university
* being unable to follow the controlled diet instructions
* being pregnant or planning to become pregnant during the study (if female)
* disorders of fat metabolism, chronic pancreatitis, had gastric bypass surgery and/or gallbladder disease
* being unable to read or communicate in English

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baranowski BJ, Oliveira BF, Falkenhain K, Little JP, Mohammad A, Beaudette SM, Finch MS, Caldwell HG, Neudorf H, MacPherson REK, Walsh JJ. Effect of exogenous beta-hydroxybutyrate on BDNF signaling, cognition, and amyloid precursor protein processing in humans with T2D and insulin-resistant rodents. Am J Physiol Cell Physiol. 2025 Feb 1;328(2):C541-C556. doi: 10.1152/ajpcell.00867.2024. Epub 2025 Jan 13. PMID 39804761

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo-Ketones: Crossover design: Placebo - washout period of >2days - Ketones
- Ketones-Placebo: Crossover design: Ketones - washout period of >2days - Placebo.
Period: Overall Study
Arm/Group | Placebo-Ketones | Ketones-Placebo
Started | 9 | 10
Completed | 8 | 10
Not Completed | 1 | 0
Not completed — not eligible | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: Total participants independent of crossover order (Placebo-Ketones and Ketones-Placebo).
Arm/Group | Overall
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 18

OUTCOME MEASURES:

1. Primary Outcome: Plasma Glucose
Description: Plasma glucose concentration after ketone or placebo ingestion
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 18 | 18
mmol/L
  Baseline | 7.3 (1.8) | 7.2 (1.8)
  30 minutes | 6.2 (1.2) | 6.6 (1.9)
  60 minutes | 6.3 (1.5) | 6.2 (1.8)
  90 minutes | 6.2 (1.5) | 5.9 (1.2)
  120 minutes | 5.7 (1.5) | 6.2 (0.9)
  150 minutes | 5.7 (1.4) | 5.7 (1.1)
  180 minutes | 5.6 (1.4) | 6.4 (1.5)

2. Secondary Outcome: Plasma Insulin
Description: Insulin across concentration after ketone or placebo ingestion
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 18 | 18
pg/mL
  baseline | 26.7 (17.4) | 28.2 (18.2)
  180minutes | 24.3 (17.2) | 21.4 (15.4)

3. Secondary Outcome: Plasma C-peptide
Description: C-peptide across concentration after ketone or placebo ingestion
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 18 | 18
pg/mL
  baseline | 4,384 (2,155) | 4,438 (2,241)
  180 minutes | 3,908 (1,859) | 3,918 (2,232)

4. Secondary Outcome: Plasma Free Fatty Acids
Description: Non-esterified fatty acid concentration after ketone or placebo ingestion
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 18 | 18
mmol/L
  baseline | 0.42 (0.14) | 0.40 (0.18)
  180 minutes | 0.18 (0.11) | 0.43 (0.16)

5. Secondary Outcome: Plasma Tumour Necrosis Factor Alpha
Description: Plasma tumour necrosis factor alpha concentration after ketone or placebo ingestion
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 18 | 18
pg/mL
  baseline | 1.1 (0.5) | 1.2 (0.4)
  180min | 1.0 (0.4) | 1.1 (0.4)

6. Secondary Outcome: Plasma Tumour Interleukin-1beta
Description: Plasma tumour interleukin-1beta concentration after ketone or placebo ingestion
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: fg/mL
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 18 | 18
fg/mL
  baseline | 253 (450) | 115 (74)
  180min | 106 (105) | 102 (41)

7. Secondary Outcome: Plasma Tumour Interleukin-6
Description: Plasma tumour interleukin-6 concentration after ketone or placebo ingestion
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 18 | 18
pg/mL
  baseline | 1.5 (0.8) | 2.7 (1.6)
  180min | 2.7 (1.6) | 2.7 (1.6)

8. Secondary Outcome: Cerebral Blood Flow
Description: Intracranial blood flow velocity measured by ultrasound
Time Frame: 180 minutes
Population: Procedure not completed due to the unavailability of a specialized research staff. Data was not and will not be obtained and reported.
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Blood Pressure
Description: Blood pressure measured manually and by Finipres
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 18 | 18
mmHg
  Systolic blood pressure baseline | 133 (18) | 130 (16)
  Systolic blood pressure 180min | 139 (19) | 136 (18)
  Diastolic blood pressure baseline | 79 (7) | 77 (10)
  Diastolic blood pressure 180min | 83 (11) | 78 (14)

10. Secondary Outcome: Cognitive Function - Digital Symbol Substitution Task
Description: Number of Correct Answers on the Digital Symbol Substitution Task. Measure of cognitive function using Brain Baseline battery on an iPad.
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 18 | 18
number correct
  baseline Digit-symbol substitution task | 32.8 (8.7) | 32.4 (8.2)
  180min Digit-symbol substitution task | 35.7 (7.5) | 34.5 (6.9)

11. Secondary Outcome: Brain-derived Neurotrophic Factor
Description: Brain-derived neurotrophic factor concentrations after ketone or placebo ingestion
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 18 | 18
ng/mL
  baseline | 7.1 (13.0) | 5.5 (8.1)
  180 minutes | 4.8 (6.7) | 5.7 (9.0)

12. Secondary Outcome: Number Blood Monocytes (x10^3 Cells/uL)
Description: Total blood monocytes count (x10^3 cells/uL) after ketone or placebo ingestion
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: x10^3 cells/uL
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 18 | 18
x10^3 cells/uL
  baseline Monocytes | 408 (171) | 442 (152)
  180min Monocytes | 445 (181) | 447 (179)

13. Secondary Outcome: Self Reported Hunger and Fullness
Description: Self reported hunger and fullness by a 0 to 100 mm Visual Analog Scale (higher scores mean greater hunger or fullness)
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 18 | 18
mm
  baseline how hungry | 46 (26) | 42 (31)
  180 minutes how hungry | 58 (21) | 60 (23)

14. Secondary Outcome: Gastrointestinal Symptoms
Description: Gastrointestinal symptom questionnaire scores after ketone or placebo ingestion on a 0 to 100 mm Visual Analog Scale (higher scores mean greater symptoms)
Time Frame: 180 minutes
Measure: Median (Full Range); unit: mm
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 18 | 18
mm
  nausea | 0 [0 to 59] | 0 [0 to 22]
  urge to vomit | 0 [0 to 32] | 0 [0 to 69]
  bloating | 0 [0 to 42] | 0 [0 to 24]
  belching | 0 [0 to 46] | 0 [0 to 59]
  cramping | 0 [0 to 12] | 0 [0 to 22]

15. Secondary Outcome: Total Energy Consumed
Description: Total energy consumed in kilocalories in buffet style meal after ketone or placebo ingestion
Time Frame: 180 minutes after ketone or placebo ingestion
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 18 | 18
kcal | 823 (377) | 948 (455)

16. Secondary Outcome: Monocyte Histone Acetylation
Description: Histone acetylation status of monocytes measured after ketone or placebo ingestion
Time Frame: 180 minutes
Population: This assay was not performed due to insufficient sample quantity.
Arm/Group | Ketone Monoester | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: About two weeks. Timeframe of first visit and second visit.
Arm/Group | Overall
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT04194450/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT04194450/SAP_001.pdf